CLINICAL TRIAL: NCT00069953
Title: A Phase II Study Of Paclitaxel-Based Chemoradiotherapy Regimen With Selective Surgical Salvage For Resectable Locoregionally Advanced Carcinoma Of The Esophagus
Brief Title: Combination Chemotherapy Followed By Chemoradiotherapy, With or Without Surgery, in Treating Patients With Resectable Locally Advanced Cancer of the Esophagus or Gastroesophageal Junction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0246; CDR0000306455
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2016-12

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage II esophageal cancer; stage III esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim; pegylated granulocyte colony-stimulating factor, human; Cisplatin; Fluorouracil; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ChemoRT and selective surgery (Experimental): Induction therapy of fluorouracil, cisplatin, paclitaxel, and pegfilgrastim OR filgrastim, then chemoradiotherapy of concurrent cisplatin and fluorouracil with external beam radiotherapy (RT), followed by selective salvage therapy.
  Interventions: Biological: filgrastim; Biological: pegfilgrastim; Drug: cisplatin; Drug: fluorouracil; Drug: paclitaxel; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — During induction therapy, patients ≤ 70 kg will receive 300 μg OR patients >70 kg will receive 480 μg subcutaneously on days 6-15 and 34-42.
  Other Names: G-CSF
Biological: pegfilgrastim — During induction therapy, patients receive 6 mg subcutaneously on days 6 and 34.
  Other Names: PEG-G-CSF
Drug: cisplatin — During induction therapy, patients receive 15 mg/m^2/day by IV over 1 hour on days 1-5 and 29-33. During radiotherapy, patients receive 15 mg/m^2/day by IV over 1 hour beginning on days 57-61.
Drug: fluorouracil — During induction therapy, patients receive 650 mg/m^2/day by IV continuously over 96 hours beginning on days 1 and 29. During radiotherapy, patients receive 300 mg/m^2/day by IV continuously over 96 hours beginning on day 57 for 5 cycles.
  Other Names: 5-FU
Drug: paclitaxel — During induction therapy, patients receive 200 mg/m^2/day by IV over 2 hours on days 1 and 29.
Procedure: conventional surgery — Patients with residual or recurrent esophageal disease 4-6 weeks after completion of chemoradiotherapy may undergo salvage esophagectomy.
Radiation: radiation therapy — External beam radiotherapy with megavoltage linear accelerators (> 6 MV) will be used to deliver multiple (> 2) field techniques. Patients will be treated 5 days/week at 1.8 Gy/day for 28 days for a total dose of 50.4 Gy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as paclitaxel, fluorouracil, and cisplatin use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells

PURPOSE: This phase II trial is studying how well combination chemotherapy followed by chemoradiotherapy, with or without surgery, works in treating patients with resectable locally advanced cancer of the esophagus or gastroesophageal junction.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of treatment with paclitaxel, cisplatin, and fluorouracil followed by chemoradiotherapy and possible surgical salvage in patients with resectable locally advanced carcinoma of the esophagus or gastroesophageal junction.
* Determine the overall and disease-free survival of patients treated with this regimen.
* Determine the treatment-related toxicity of this regimen in these patients.
* Determine the tolerance to surgical salvage in patients treated with this regimen.
* Determine the morbidity and mortality of surgical salvage in patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive fluorouracil (5-FU) IV continuously over 96 hours beginning on days 1 and 29; cisplatin IV over 1 hour on days 1-5 and 29-33; paclitaxel IV over 2 hours on days 1 and 29; and pegfilgrastim subcutaneously (SC) on days 6 and 34 OR filgrastim (G-CSF) SC on days 6-15 and 34-42. Treatment continues in the absence of unacceptable toxicity.
* Chemoradiotherapy: Patients receive cisplatin IV over 1 hour on days 57-61 and 5-FU IV continuously on days 57-61, 64-68, 71-75, 78-82, 85-89, and 92-96. Patients concurrently undergo external beam radiotherapy on days 57-61, 64-68, 71-75, 78-82, 85-89, and 92-96.

Patients with residual or recurrent esophageal disease 4-6 weeks after completion of chemoradiotherapy may undergo salvage esophagectomy.

Patients are followed periodically.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma or adenocarcinoma of the esophagus or gastroesophageal junction

  * Primary (non-recurrent) disease
  * Amenable to resection
  * Stage greater than T1, N0 by endoscopic ultrasound
  * Must be entirely confined to the esophagus or gastroesophageal junction and periesophageal soft tissue
  * Tumor may not extend more than 2 cm into the stomach
* No multiple primary carcinomas of the esophagus
* No cervical esophageal carcinoma or tumors less than 5 cm from cricopharyngeus
* No evidence of disseminated cancer

  * Suggestion of liver metastases by positron emission tomography must be proven negative by biopsy or other imaging studies
  * Palpable supraclavicular nodes must be negative for cancer by biopsy
* Bronchoscopy required for lesions less than 26 cm from the incisors to exclude tracheoesophageal fistula or invasion
* No celiac adenopathy greater than 2 cm

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 150,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Not specified

Renal

* Creatinine no greater than 1.5 mg/dL AND/OR
* Creatinine clearance at least 65 mL/min
* Calcium no greater than 11 mg/dL

Cardiovascular

* No uncontrolled heart disease
* No uncontrolled hypertension

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to comprehend study requirements and considered likely to comply with study parameters
* No other malignancy within the past 5 years except curable nonmelanoma skin cancer or carcinoma in situ of the cervix
* No uncontrolled diabetes
* No hypersensitivity to E. coli-derived products

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 5 years since prior systemic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior chest or upper abdomen radiotherapy

Surgery

* No prior esophageal or gastric surgery

Other

* No concurrent photodynamic therapy
* No other concurrent investigational agents for esophageal carcinoma

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2003-09; Primary Completion 2007-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G. Swisher, MD, Study Chair — M.D. Anderson Cancer Center
Locations (97):
- United States (97):
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Saint Rose Hospital, Hayward, California
  - Providence Holy Cross Cancer Center, Mission Hills, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Summit Medical Center, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - J.C. Robinson, M.D. Regional Cancer Center, San Pablo, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Hospital of Saint Raphael, New Haven, Connecticut
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Ochsner Clinic of Baton Rouge, Baton Rouge, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Foote Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Hattiesburg Clinic, P.A., Hattiesburg, Mississippi
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Marlton, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Community Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Albuquerque Regional Medical Center at Lovelace Sandia Health System, Albuquerque, New Mexico
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilmed Radiation Oncology Services, Wilson, North Carolina
  - Akron City Hospital, Akron, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Result] Swisher SG, Winter KA, Komaki RU, Ajani JA, Wu TT, Hofstetter WL, Konski AA, Willett CG. A Phase II study of a paclitaxel-based chemoradiation regimen with selective surgical salvage for resectable locoregionally advanced esophageal cancer: initial reporting of RTOG 0246. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):1967-72. doi: 10.1016/j.ijrobp.2011.01.043. Epub 2011 Apr 18. PMID 21507583

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ChemoRT and Selective Surgery
Started | 43
Completed | 41 (Subjects with data available for the primary analysis are considered to have completed the study)
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: All eligible patients.
Arm/Group | ChemoRT and Selective Surgery
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: years] | 59 [42 to 81]
Gender [Count of Participants; unit: Participants]
  Female | 7
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (1-year Rate Reported)
Description: One-year survival estimate is reported. Survival time is defined as time from registration to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at date of last contact. This analysis was planned to occur when all patients had been potentially followed for 1 year. On the basis of a 1-year survival rate of 60% from the Radiation Therapy Oncology Group (RTOG) esophageal database, 38 analyzable patients with a 1-year survival rate of 77.5% or better was needed for this trial to be deemed promising enough for development of a Phase III protocol (type I error of 0.05 and type II error of 0.20).
Time Frame: From registration to date of death or last follow-up. Analysis occurs after all patients have been potentially followed for 1 year.
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ChemoRT and Selective Surgery
Number analyzed (Participants) | 41
percentage of participants | 71 [54 to 82]

2. Secondary Outcome: Frequency of Major (Grade 4) Acute Treatment-related Toxicities
Time Frame: From start of chemotherapy to surgery or 2 months after chemoradiation (for patients not undergoing surgery).
Reporting Status: Not Posted

3. Secondary Outcome: Frequency of Patients With Persistent or Recurrent Disease Eligible for Surgical Salvage Resection
Time Frame: Analysis occurs with the primary outcome measure.
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-serious adverse events (AE). Data is reported for all registered patients.
Arm/Group | ChemoRT and Selective Surgery
Serious Adverse Events (participants affected / at risk) | 26/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ChemoRT and Selective Surgery (N=41)
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 1
Arrhythmia NOS (Cardiac disorders) | 1
Diarrhea NOS (Gastrointestinal disorders) | 4
Esophageal spasm (Gastrointestinal disorders) | 5
Esophagitis NOS (Gastrointestinal disorders) | 2
GI-other (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Tracheo-oesophageal fistula NOS (Gastrointestinal disorders) | 1
Vomiting NOS (Gastrointestinal disorders) | 4
Chest pain (General disorders) | 2
Pain due to radiation (General disorders) | 3
Pain-other (General disorders) | 3
Infection NOS (Infections and infestations) | 2
Infection, Other (Infections and infestations) | 1
Neutropenia (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia NOS (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 1
Dizziness (exc vertigo) (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Renal failure NOS (Renal and urinary disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Late RT Toxicity: Lung: NOS (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 2
Thrombosis NOS (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ChemoRT and Selective Surgery (N=41)
Hemoglobin decreased (Blood and lymphatic system disorders) | 36
Constipation (Gastrointestinal disorders) | 18
Diarrhea NOS (Gastrointestinal disorders) | 16
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 7
Esophageal spasm (Gastrointestinal disorders) | 11
Esophagitis NOS (Gastrointestinal disorders) | 15
GI-other (Gastrointestinal disorders) | 9
Late RT Toxicity: Esophagus: NOS (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 29
Stomatitis (Gastrointestinal disorders) | 8
Vomiting NOS (Gastrointestinal disorders) | 18
Chest pain (General disorders) | 3
Fatigue (General disorders) | 37
Pain due to radiation (General disorders) | 6
Pain-other (General disorders) | 11
Pyrexia (General disorders) | 4
Infection NOS (Infections and infestations) | 4
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 12
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 6
Blood alkaline phosphatase NOS increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 4
Blood creatinine increased (Investigations) | 5
Leukopenia NOS (Investigations) | 28
Lymphopenia (Investigations) | 7
Metabolic-Other (Investigations) | 3
Neutropenia (Investigations) | 14
Platelet count decreased (Investigations) | 24
Weight decreased (Investigations) | 19
Anorexia (Metabolism and nutrition disorders) | 22
Blood albumin decreased (Metabolism and nutrition disorders) | 7
Blood magnesium decreased (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 7
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia NOS (Metabolism and nutrition disorders) | 25
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypoglycaemia NOS (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 14
Dizziness (exc vertigo) (Nervous system disorders) | 8
Headache NOS (Nervous system disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 23
Taste disturbance (Nervous system disorders) | 9
Insomnia NEC (Psychiatric disorders) | 10
Renal/GU-Other (Renal and urinary disorders) | 3
Urinary frequency (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 24
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 9
Localized exfoliation (Skin and subcutaneous tissue disorders) | 4
Hypotension NOS (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.